CLINICAL TRIAL: NCT01717014
Title: Evaluating the Radial Reload Stapler With Tri-Staple TM Technology During Open Low Anterior Resection for Rectal Cancer: A Prospective Multicenter Case Series
Brief Title: Radial Reload Open LAR Case Series
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Collaborators: Duke University (Other); Providence Medical Research Center (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVLARO0286
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Low Anterior Resection; Proctosigmoid Resection; Rectal Cancer
Keywords: rectal cancer; stapler
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Covidien Radial Reload Stapler with Tri-Staple Technology (Experimental): Covidien Radial Reload Stapler with Tri-Staple Technology in open low anterior resection or anterior proctosigmoidectomy
  Interventions: Device: Covidien Radial Reload Stapler with Tri-Staple Technology

INTERVENTIONS:
Device: Covidien Radial Reload Stapler with Tri-Staple Technology — Case series of patients already selected to undergo an open LAR or proctosigmoidectomy using the Radial Reload Stapler

SUMMARY:
The purpose of this research study is to evaluate the safety and feasibility of the Radial Reload Stapler during open LAR for rectal cancer. The surgeon will complete questionnaires relating to the function of the device.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to understand and sign Informed Consent Form.
2. The subject is between 18-85 years of age.
3. The subject is anticipated to undergo a resection of the rectum with anastomosis below the peritoneal reflection for the treatment of rectal cancer.
4. The subject is anticipated to undergo mobilization and stapling of the rectum through an open incision.

Exclusion Criteria:

1. Any female patient, who is pregnant, suspected pregnant, or nursing.
2. The participant is unable or unwilling to comply with the study requirements, follow-up schedule.
3. The participant has co-morbidities which, in the opinion of the investigator, will not be appropriate for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of South Florida, Tampa, Florida
  - Duke University, Durham, North Carolina
  - Providence Medical Center, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters] | 175.1 (4.3)
Weight [Mean (Standard Deviation); unit: kilograms] | 88.7 (18.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.0 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Staple Line
Description: The surgeons ability to achieve a staple line at the desired level of the rectum.
Time Frame: Operative
Measure: Number; unit: participants
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
participants | 7

2. Primary Outcome: Distal Margins
Description: The ability to achieve adequate distal margins (defined as >2cm [or >1cm with clear histologic evaluation]) in the low rectum.
Time Frame: Operative
Measure: Number; unit: participants
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
participants | 8

3. Secondary Outcome: Usability: Visibility
Description: Visibility measured by surgeon usability questionnaire.
Time Frame: Operatively
Measure: Number; unit: % of cases surgeon agree/strongly agree
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
% of cases surgeon agree/strongly agree
  Visibility adequate when RR was used operatively | 100
  Did instrument impede visibility | 0

4. Secondary Outcome: Usability: Access
Description: Access measured by surgeon usability questionnaire
Time Frame: Operatively
Measure: Number; unit: % of cases surgeon agree/strongly agree
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
% of cases surgeon agree/strongly agree
  Radial Reload (RR) easy to place in pelvis | 100
  RR was able to get low in pelvis | 100
  RR was easy to place in the colon & rectum | 100
  Was rectum contained in the device after clamping | 12.5
  RR retained an adequate tissue during clamping | 100
  Was the rectum transected in one firing | 12.5

5. Secondary Outcome: Usability: Manueverability
Description: Manueverability measured by surgeon usability questionnaire. Question: Maneuverability of Radial reload during the procedure was adequate
Time Frame: Operatively
Measure: Number; unit: % of cases surgeon agree/strongly agree
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Number analyzed (Participants) | 8
% of cases surgeon agree/strongly agree | 87.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 30 day follow-up visit
Arm/Group | Covidien Radial Reload Stapler With Tri-Staple Technology
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Covidien Radial Reload Stapler With Tri-Staple Technology (N=8)
Ileus (Gastrointestinal disorders) | 2 (2)
Pelvic abscess (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Covidien Radial Reload Stapler With Tri-Staple Technology (N=8)
Urinary retention (Renal and urinary disorders) | 1 (1)
Post-operative ileus (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No